CLINICAL TRIAL: NCT06342284
Title: Patient-Generated Health Data Collection During Chemoradiotherapy for Lung Cancer: A Pilot Study
Brief Title: Patient-Generated Health Data Collection During Chemoradiotherapy for Lung Cancer
Acronym: PGHD
Status: Recruiting | Type: Observational
Sponsor: The New York Proton Center (Other)
Responsible Party: Sponsor
Other Study IDs: NYPC ERC# 2021-030
Record Dates: First submitted 2024-03-20; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Thoracic Cancer

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Proton Beam Radiation with or without concurrent chemotherapy — Curative-intent fractionated proton beam thoracic radiotherapy, with or without concurrent chemotherapy

SUMMARY:
This is an observational study involving the collection of patient-generated health data using an Apple Watch, a home pulse oximeter, and a smartphone during a course of proton beam radiotherapy for lung cancer. The study period over which this information is collected will range from the day of study enrollment until two weeks after radiotherapy completion. Subjects will complete a short satisfaction survey at the end of the study period. Other information that is collected as part of routine care for this patient population will be extracted from subjects' medical records during the study period and afterwards.

DETAILED DESCRIPTION:
This is an observational study involving the collection of patient-generated health data using an Apple Watch, a home pulse oximeter, and a smartphone during a course of proton beam radiotherapy for lung cancer. The study period over which this information is collected will range from the day of study enrollment until two weeks after radiotherapy completion. Subjects will complete a short satisfaction survey at the end of the study period. Other information that is collected as part of routine care for this patient population will be extracted from subjects' medical records during the study period and afterwards.

Primary Objective

• To demonstrate the feasibility of patient-generated health data collection during thoracic proton beam radiotherapy for lung cancer.

Secondary Objective • To demonstrate the face validity of physical activity and vital sign data collected during proton beam radiotherapy for lung cancer.

Exploratory Objective

• To explore associations between radiotherapy treatment parameters, wearable device data, patient-reported outcomes, adverse events, and long-term clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Plan for fractionated (≥15 treatments) proton beam thoracic radiotherapy with curative intent for lung cancer
* Non-small cell lung cancer (NSCLC) or small cell lung cancer (SCLC) histology is permitted.
* Concurrent chemotherapy is permitted but not required..
* Previous thoracic radiotherapy is allowed.
* Ability to complete study surveys in English or Spanish
* Age >/= 18
* Concurrent enrollment on other trials is permitted
* Patients who already use wearable devices and/or smartphones that monitor physical activity are eligible for this trial, provided they agree to utilize the devices provided by the study team during the study period
* All patients must sign study-specific informed consent prior to study entry

Exclusion Criteria:

* Ongoing treatment for another cancer that is expected to affect the toxicity profile of thoracic radiotherapy
* Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 17 years old that will be receiving proton beam thoracic radiotherapy with curative intent for lung cancer.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-03-22 (Actual); Primary Completion 2026-03-21 (Estimated); Study Completion 2031-03-21 (Estimated)

PRIMARY OUTCOMES:
Demonstrate the feasibility of patient-generated health data collection during thoracic proton beam radiotherapy for lung cancer, based on the quantity of data collected from the day of radiotherapy initiation to the day of radiotherapy completion. | 4-5 Weeks
  Feasibility assessed based on the quantity of data collected from day of radiotherapy initiation to day of radiotherapy completion. The feasibility of physical activity data collection will be assessed based on usage information provided by the Apple Watch. Descriptive statistics to be used to report the distribution of average use times in the study cohort and the proportion of days subjects wear the Apple Watch for at least 8 hours. The feasibility of daily home pulse oximeter data collection reported using frequencies and percentages. The feasibility of weekly electronic PRO collection reported using frequencies and percentages.

SECONDARY OUTCOMES:
Demonstrate the face validity of physical activity and vital sign data collected in this trial by reviewing the distribution of values obtained for each measure quantitatively using descriptive statistics. | 4-5 Weeks
  Face validity will be evaluated by reviewing the distribution of values obtained for each measure quantitatively using descriptive statistics (mean, standard deviation, median, range) and visually using histograms and boxplots. Additionally, the proportion of reported measures outside of the expected range based on subjects' medical conditions and data obtained during clinic visits (i.e., non-physiologic outliers) will be estimated by the study team. Data elements will be deemed to have face validity if less than 5% of the collected values fall outside the expected range.

OTHER OUTCOMES:
Assess associations between radiotherapy treatment parameters, wearable device data, patient-reported outcomes, adverse events, and long-term clinical outcomes using inferential statistical analyses. | 5 Years
  Inferential statistical analyses carried out in support of this objective will be exploratory, recognizing the feasibility nature of the study, the associated lack of statistical power, and that these analyses are intended to estimate effect sizes to inform future studies.

CONTACTS AND LOCATIONS:
Overall Officials: Nitin Ohri, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- New York Proton Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data planned to be shared